CLINICAL TRIAL: NCT05176548
Title: Registry of Patients with Suspected Amyloidosis in Heart Failure: Regamic
Brief Title: Registry of Patients with Suspected Amyloidosis in Heart Failure
Acronym: Regamic
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: REGAMIC-1450-N-21
Record Dates: First submitted 2021-11-08; First posted 2022-01-04 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
Keywords: Amyloidosis
MeSH Terms: conditions — Heart Failure; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients in whom Cardiac Amyloidosis is confirmed
  Interventions: Diagnostic Test: Bone-cardiac scintigraphy
- Group 2: Patients in whom Cardiac Amyloidosis is ruled out
  Interventions: Diagnostic Test: Bone-cardiac scintigraphy

INTERVENTIONS:
Diagnostic Test: Bone-cardiac scintigraphy — Patients with confirmed ATTR type CA will undergo a study of mutations in the TTR gene
  Other Names: Laboratory test to rule out monoclonal protein

SUMMARY:
Observational multicenter registry of cohorts with follow-up.

Patients with heart failure, age ≥ 18 years, with clinical suspicion of cardiac amyloidosis and any LVEF value, treated in the field of Internal Medicine.

Initially, a duration of two years was established to recruit at least 150 patients in the group with AC, and a follow-up of two years.

Upon completion of the two years of follow-up, the continuity or completion of the registry will be assessed.

DETAILED DESCRIPTION:
Observational, cohort study with a duration of two years to recruit at least 150 patients in the group with CA, and a follow-up of two years. The investigators estimate a sample size of at least 150 patients in the Group 1 (CA confirmed), and a total of 450 patients.

The primary objectives of this study are:

* To evaluate differential characteristics between two groups of patients with Heart

Failure with clinical suspicion of Cardiac Amyloidosis (CA):

* Group 1: Patients in whom CA is confirmed.
* Group 2: Patients in whom CA is ruled out.

  * Clinical, laboratory, electrocardiographic, echocardiographic characteristics, and other studies (MRI, biopsies, etc.) will be compared between both groups.

The secondary objectives are:

* To evaluate the clinical and complementary test data on which the suspicion of the diagnosis of AC has been based.
* To identify prognostic differences between both groups by comparing readmission rates, mortality and other events of patients with CA and without CA in a period of two years.

The patients included in the study are elderly patients, of both genders, with heart failure, who have undergone an echocardiogram in the last 24 months, with a clinical suspicion of amyloidosis.

All patients who meet inclusion criteria will be included from January 2022 to December 2023.

The following studies are performed on each patient:

* Clinical, laboratory, electrocardiographic, echocardiographic.
* Bone-cardiac scintigraphy.
* Laboratory test to rule out monoclonal protein.
* The number of readmissions, emergency room visits, and mortality in the 24 months following their inclusion will be recorded.

A descriptive analysis of the data and a comparative analysis will be made in relation to different variables. The association of different variables with readmission and mortality data will be assessed using univariate and multivariate analysis. An analysis of survival curves will also be performed using the Kaplan-Meier method using the log-rank test.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age ≥ 18 years.
* Both genders.
* Heart Failure (2021 European Society of Cardiology criteria)
* Any LVEF value.
* Outpatients or hospitalized patients in Internal Medicine Units
* Patients with suspicion criteria proposed by the European Society of Cardiology:

  * Ventricular hypertrophy ≥ 12 mm

And one or more of the following criteria:

* Heart failure in ≥ 65 years
* Aortic stenosis in ≥ 65 years
* Hypotension or Normotensive if previously hypertensive
* Sensory involvement, autonomic dysfunction
* Peripheral polyneuropathy
* Proteinuria
* Skin bruising (eg, periorbital purpura)
* Bilateral carpal tunnel syndrome
* Ruptured biceps tendon
* In CMR: Subendocardial / transmural late gadolinium enhancement (LGE), or increased extracellular volume (ECV)
* In ECO: Reduced longitudinal strain with apical sparing
* Reduced QRS voltage to mass ratio
* Pseudo Q waves on ECG
* Atrioventricular conduction disease
* Possible family history of ATTRv

EXCLUSION CRITERIA:

* Refusal to participate in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnostic Test: Bone-cardiac scintigraphy with Tc-DPD (or similar: Tc-PYP or Tc-HMDP) to evaluate the degree of cardiac uptake from 0 to 3 degrees.
  Diagnostic Test: Proteinogram and serum immunoglobulins. Light chains free in serum -Freelite-. Immunofixation in serum and urine Analysis to rule out the presence of monoclonal protein in blood and urine.
  Patients with confirmed ATTR type Cardiac Amyloidosis will undergo a study of mutations in the TTR gene
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differential characteristics between two groups | Up to two years
  Number of biopsies performed between both groups.

SECONDARY OUTCOMES:
Prognostic differences between both groups | Up to two years
  Readmission rate of patients with AC and without AC in a period of two years.
Prognostic differences between two groups | Up to Two years
  Mortality rate of patients with AC and without AC in a period of two years.

CONTACTS AND LOCATIONS:
Overall Officials: Prado Salamanca-Bautista, MD, PhD, Principal Investigator — Hospital Universitario Virgen Macarena; Rocio Ruiz-Hueso, MD, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, SEVILLA, Spain

IPD SHARING:
Plan to Share IPD: No